CLINICAL TRIAL: NCT00202397
Title: Phase 2 Study of Riluzole Effects on Patients With Chronic Cerebellar Ataxia
Brief Title: Effect of Riluzole as a Symptomatic Approach in Patients With Chronic Cerebellar Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: S. Andrea Hospital (Other)
Responsible Party: Principal Investigator, Giovanni Ristori, MD, PhD, S. Andrea Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEU - RLZ - 05
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Hereditary Ataxia; Multiple Sclerosis; Cerebellar Ataxia
Keywords: cerebellar ataxia; deep cerebellar nuclei (DCN); small-conductance calcium-activated potassium(SK)channels; riluzole; Sporadic ataxia; Multiple system atrophy type C
MeSH Terms: conditions — Spinocerebellar Degenerations; Multiple Sclerosis; Cerebellar Ataxia | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Placebo Comparator): placebo bid for 8 weeks
  Interventions: Other: placebo
- 1 (Experimental): Riluzole, capsule-shaped 50 mg tablets bid for 8 weeks
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole — capsule-shaped 50 mg tablets bid for 8 weeks
  Other Names: Rilutek ATC Code N07X X02
  Arms: 1
Other: placebo — capsule-shaped tablet bid for 8 weeks
  Arms: 2

SUMMARY:
Cerebellar disorders are often disabling and symptomatic therapies are limited to few options that are partially effective. It seems therefore appropriate to search for additional approaches.

Purkinje cells are the sole output of the cerebellar cortex: they project inhibitory signals to the deep cerebellar nuclei (DCN), which have a critical role in cerebellar function and motor performance. DCN neurons fire spontaneously in the absence of synaptic input from Purkinje neurons and modulation of the DCN response by Purkinje input is believed to be responsible for coordination of movement. Recent evidences support the notion that an increase in DCN excitability may be an important step in the development of cerebellar ataxia and point to the underlying molecular mechanisms: the inhibition of small-conductance calcium-activated potassium (SK) channels, that causes an increase of the firing frequency in DCN, correlates with cerebellar ataxia.

The rationale of the present project is that SK channel openers, such as riluzole, may have a beneficial effect on cerebellar ataxia.

The researchers propose to perform a pilot study investigating safety and efficacy of riluzole, an approved treatment for amyotrophic lateral sclerosis, as a symptomatic approach in patients with chronic cerebellar ataxia.

DETAILED DESCRIPTION:
Forty patients with chronic cerebellar ataxia will be enrolled in a double-bind, randomized, placebo-controlled trial.

By central randomisation, patients will take 50 mg of riluzole or placebo twice daily for 8 weeks.

Electrocardiogram routine laboratory tests and pregnancy tests will be performed before drug administration, after 4 weeks of treatment and at the end of the study (after 8 weeks of treatment).

At the same time points the International Cooperative Ataxia Rating Scale (ICARS) for pharmacological assessment of the cerebellar syndrome will be administered to the two groups (riluzole and placebo) of patients. To guarantee the evaluation of the results in blind conditions, the neurologists who will evaluate the ICARS scores will be different from those who will deal with randomisation and follow-up of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cerebellar degeneration (heredoataxias, sporadic idiopathic ataxia, multiple system atrophy type C)
* Patients who meet McDonald criteria for probable or definite multiple sclerosis (MS) with chronic cerebellar ataxia (not acute cerebellar ataxia due to relapse)
* Age between 18 and 80 years

Exclusion Criteria:

* Ataxia due to other diseases
* Acute cerebellar ataxia
* Use of other drugs for chronic ataxia
* Serious concomitant illnesses (cardiac arrhythmias, haematological and hepatic diseases)
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The International Cooperative Ataxia Rating Scale (ICARS) total scores and subscores (oculomotor, kinetic, postural, speech), comparing the three time points in the treated versus placebo group | pre-treatment, after 4 weeks of treatment and at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Marco Salvetti, Assoc. Prof, Study Director — S.Andrea Hospital, University of Rome "La Sapienza"; Giovanni Ristori, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- S.Andrea Hospital - University of Rome "La Sapienza", Rome, Italy

REFERENCES:
- [Background] Shakkottai VG, Chou CH, Oddo S, Sailer CA, Knaus HG, Gutman GA, Barish ME, LaFerla FM, Chandy KG. Enhanced neuronal excitability in the absence of neurodegeneration induces cerebellar ataxia. J Clin Invest. 2004 Feb;113(4):582-90. doi: 10.1172/JCI20216. PMID 14966567
- [Background] Aizenman CD, Huang EJ, Linden DJ. Morphological correlates of intrinsic electrical excitability in neurons of the deep cerebellar nuclei. J Neurophysiol. 2003 Apr;89(4):1738-47. doi: 10.1152/jn.01043.2002. PMID 12686564
- [Background] Raman IM, Gustafson AE, Padgett D. Ionic currents and spontaneous firing in neurons isolated from the cerebellar nuclei. J Neurosci. 2000 Dec 15;20(24):9004-16. doi: 10.1523/JNEUROSCI.20-24-09004.2000. PMID 11124976
- [Background] Cao YJ, Dreixler JC, Couey JJ, Houamed KM. Modulation of recombinant and native neuronal SK channels by the neuroprotective drug riluzole. Eur J Pharmacol. 2002 Aug 2;449(1-2):47-54. doi: 10.1016/s0014-2999(02)01987-8. PMID 12163105
- [Background] Doble A. The pharmacology and mechanism of action of riluzole. Neurology. 1996 Dec;47(6 Suppl 4):S233-41. doi: 10.1212/wnl.47.6_suppl_4.233s. PMID 8959995
- [Background] Trouillas P, Takayanagi T, Hallett M, Currier RD, Subramony SH, Wessel K, Bryer A, Diener HC, Massaquoi S, Gomez CM, Coutinho P, Ben Hamida M, Campanella G, Filla A, Schut L, Timann D, Honnorat J, Nighoghossian N, Manyam B. International Cooperative Ataxia Rating Scale for pharmacological assessment of the cerebellar syndrome. The Ataxia Neuropharmacology Committee of the World Federation of Neurology. J Neurol Sci. 1997 Feb 12;145(2):205-11. doi: 10.1016/s0022-510x(96)00231-6. PMID 9094050
- See also: sponsor site — http://www.ospedalesantandrea.it